CLINICAL TRIAL: NCT01195467
Title: A Phase III, Open-label, Single Centre, Single-arm, Pilot Study to Assess the Feasibility of Switching, Individuals Receiving Efavirenz With Continuing Central Nervous System (CNS) Toxicity, to Raltegravir
Brief Title: Atripla to Raltegravir Switch Study for CNS Toxicity
Acronym: SSAT036
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSAT 036
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Results first posted 2014-11-04 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Raltegravir Potassium; Emtricitabine; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Subjects Truvada/Raltegravir (Experimental): All Subjects will receive the same intervention, Truvada/Raltegravir
  Interventions: Drug: Truvada/Raltegravir

INTERVENTIONS:
Drug: Truvada/Raltegravir — All subjects currently on Atripla® will switch to Truvada/Raltegravir
  Other Names: Truvada® = tenofovir + emtricitabine; Atripla® = tenofovir + emtricitabine + efavirenz; Raltegravir = isentress

SUMMARY:
The purpose of the study is to investigate the benefits of switching away from efavirenz (part of the combination pill, Atripla®) in patients with central nervous system side effects (such as insomnia {difficulty with sleeping}, bad dreams etc). The investigators will investigate the effect of switching to Truvada (a combination pill of tenofovir and emtricitabine, the other two components of Atripla) plus raltegravir.

Raltegravir is a licensed drug for HIV treatment which showed side effects were fewer in number when compared to efavirenz in 2 other clinical studies, where patients were starting HIV treatment for the first time.

This study will also investigate the safety (in terms of other side effects and the routine blood tests which the investigators ordinarily use to monitor your treatment) and monitor effectiveness, your viral load and CD4 counts, when you switch treatment from Atripla® to Truvada/raltegravir.

DETAILED DESCRIPTION:
The majority of individuals who commence treatment for HIV in the UK start with a regimen that includes EFV in combination with other antiretrovirals. These regimens are convenient (once daily dosing) and highly efficacious. However EFV has several potential drawbacks including continued CNS toxicity, the potential for teratogenesis and a low barrier to the development of virological resistance.

Clinically controlled trials frequently reported undesirable nervous system side effects in patients receiving 600 mg EFV with other antiretroviral agents, including dizziness, insomnia, somnolence, impaired concentration and abnormal dreaming. CNS symptoms of moderate to severe intensity were experienced by 19.4% of patients compared to 9.0% of patients receiving control regimens. These symptoms were severe in 2.0% of patients receiving EFV 600 mg daily and in 1.3% of patients receiving control regimens. In clinical studies 2.1% of patients treated with 600 mg of EFV discontinued therapy because of nervous system symptoms

The majority of individuals who commence treatment for HIV in the UK start with a regimen that includes EFV in combination with other antiretrovirals. These regimens are convenient (once daily dosing) and highly efficacious. However EFV has several potential drawbacks including continued CNS toxicity, the potential for teratogenesis and a low barrier to the development of virological resistance.

Clinically controlled trials frequently reported undesirable nervous system side effects in patients receiving 600 mg EFV with other antiretroviral agents, including dizziness, insomnia, somnolence, impaired concentration and abnormal dreaming. CNS symptoms of moderate to severe intensity were experienced by 19.4% of patients compared to 9.0% of patients receiving control regimens. These symptoms were severe in 2.0% of patients receiving EFV 600 mg daily and in 1.3% of patients receiving control regimens. In clinical studies 2.1% of patients treated with 600 mg of EFV discontinued therapy because of nervous system symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. is male or female aged 18 years or above
2. has a documented HIV-1 infection
3. has signed the Informed Consent Form voluntarily
4. is willing to comply with the protocol requirements
5. has an HIV-plasma viral load at screening <50 copies/mL
6. has a CD4 cell count at Screening >50 cells/mm3
7. has been on a stable ART, with at least 3 licensed agents, one of which being EFV, for at least 12 weeks at Screening, and has been on Atripla for at least 4 weeks at screening; the subject must be willing to stay on treatment until Baseline
8. estimated glomerular filtration rate (by MDRD or CG methods) >50 ml/min.
9. has symptomatic toxicity associated with EFV after at least 12 weeks of therapy
10. if female and of childbearing potential, she is using effective birth control methods (as agreed by the investigator) and is willing to continue practising these birth control methods during the trial and for at least 30 days after the end of the trial (or after last intake of investigational ARVs); Note: Women who are postmenopausal for least 2 years, women with total hysterectomy, and women who have a tubal ligation are considered of non-childbearing potential
11. if a heterosexually active male, he is using effective birth control methods and is willing to continue practising these birth control methods during the trial and until follow-up visit

Exclusion Criteria:

1. is infected with HIV-2
2. is using any concomitant therapy disallowed as per SPC for the study drugs (section 5.2)
3. has a currently active AIDS defining illness (Category C conditions according to the CDC Classification System for HIV Infection 1993) with the following exceptions (must be discussed with the sponsor prior to enrolment):

   * Stable cutaneous Kaposi's Sarcoma (no pulmonary or gastrointestinal involvement other than oral lesions) unlikely to require systemic therapy during the trial period
   * CD4 count less than 200 cells/mm3 Note: Primary and secondary prophylaxis for an AIDS defining illness is allowed
4. has acute viral hepatitis including, but not limited to, A, B, or C
5. has chronic hepatitis B and/or C with AST and/or ALT >5 x ULN Note: Subjects co-infected with chronic HBV or HCV can enter the trial if clinically stable and not expected to require treatment during the trial period.
6. has received any investigational drug within 30 days prior to the trial drug administration
7. Prior exposure to raltegravir or investigational integrase inhibitors
8. Any tenofovir or emtricitabine associated resistance mutations
9. No baseline resistance test available
10. Clinically significant allergy or hypersensitivity to any trial medication excipients
11. If female, she is pregnant or breastfeeding
12. screening blood results with any grade 3 / 4 toxicity according to Division of AIDS (DAIDS) grading scale, except: asymptomatic grade 3 glucose, amylase or lipid elevation or asymptomatic grade 4 triglyceride elevation (re-test allowed).
13. Clinical or laboratory evidence of significantly decreased hepatic function or decompensation: INR > 1.5 or albumin < 30g/L or bilirubin > 2.5 x ULN
14. Resolution of their CNS toxicity between Screening and Baseline visits
15. Any condition (including drug/alcohol abuse) or laboratory results which, in the investigator's opinion, interfere with assessments or completion of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Nelson, Dr, Principal Investigator — St Stephen's AIDS Trust
Locations (1):
- St Stephen's Centre, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: No randomisation as this is a single arm trial. All subjects switched from one tablet once daily of Atripla to Truvada at baseline and trested for 12 weeks.
Period: Overall Study
Arm/Group | Single Arm
Started | 40
Completed | 30
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 38
Region of Enrollment [Number; unit: participants]
  United Kingdom | 40

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Neuropsychiatric and Central Nervous System (CNS) Toxicity of Raltegravir Therapy After 4 Weeks on Treatment
Description: To assess the rate of neuropsychiatric and central nervous system (CNS) toxicity as measured from baseline to 4 weeks of raltegravir therapy as measured by sleep questionnaire & CNS toxicity (as determined by questionnaire based on efavirenz SPC and graded based on the ACTG adverse event scale)
Time Frame: 4 weeks
Measure: Number; unit: percentage improvement in CNS score
Groups:
- Single Arm: No randomisation as this is a single arm trial. All subjects switched from one tablet once daily of Atripla to Truvada at baseline and treated for 12 weeks.
Arm/Group | Single Arm
Number analyzed (Participants) | 40
percentage improvement in CNS score | 26

2. Secondary Outcome: The Rate of Neuropsychiatric and Central Nervous System (CNS) Toxicity of Raltegravir Therapy After 12 Weeks on Treatment
Description: The rate of neuropsychiatric and central nervous system (CNS) toxicity as measured after 12 weeks of raltegravir therapy as measured by :
  * Sleep questionnaire
  * CNS toxicity (as determined by questionnaire based on efavirenz SPC and graded based on the ACTG adverse event scale)
Time Frame: baseline to week 12
Measure: Number; unit: percentage of improvement in sleep score
Arm/Group | Single Arm
Number analyzed (Participants) | 40
percentage of improvement in sleep score | 25

3. Secondary Outcome: Change From Baseline to Week 12 in CD4+ Count After 12 Weeks of Raltegravir
Description: Change from baseline to week 12 in CD4+ count after 12 weeks of raltegravir having switched from efavirenz-containing therapy
Time Frame: baseline to week 12
Reporting Status: Not Posted

4. Secondary Outcome: Proportion of Patients With Viral Load < 50 Copies/mL and <400 Copies/ml at Weeks 4 and 12 After Switching to Raltegravir
Description: To assess the proportion of patients with viral load < 50 copies/mL and <400 copies/ml at weeks 4 and 12 after switching to raltegravir
Time Frame: week 4 to week 12
Reporting Status: Not Posted

5. Secondary Outcome: Change in Fasting Lipids (Total Cholesterol and Subfractions and Triglycerides) After 4 and 12 Weeks of Raltegravir
Description: To assess the change in fasting lipids (total cholesterol and subfractions and triglycerides) after 4 and 12 weeks of raltegravir
Time Frame: week 4 to week 12
Reporting Status: Not Posted

6. Secondary Outcome: Proportion of Patients With Grade 2-4 Laboratory Parameters (Excluding Lipids) After 12 Weeks of Raltegravir Compared With Baseline
Description: To assess the proportion of patients with grade 2-4 laboratory parameters (excluding lipids) after 12 weeks of raltegravir compared with baseline
Time Frame: baseline to week 12
Reporting Status: Not Posted

7. Secondary Outcome: Proportion of Patients With Grade 2-4 Non-CNS Adverse Events After 12 Weeks of Raltegravir Compared With Baseline
Description: To assess the proportion of patients with grade 2-4 non-CNS adverse events after 12 weeks of raltegravir compared with baseline
Time Frame: baseline to week 12
Reporting Status: Not Posted

8. Secondary Outcome: Change From Baseline in Adherence From Baseline After 12 Weeks of Raltegravir as Measured by the Adherence Questionnaire: Medication Adherence Self-Report Inventory (M-MASRI)
Description: To assess the change from baseline in adherence from baseline after 12 weeks of raltegravir as measured by the adherence questionnaire: Medication Adherence Self-Report Inventory (M-MASRI)
Time Frame: baseline to week 12
Reporting Status: Not Posted

9. Secondary Outcome: Change From Baseline of CNS Toxicity as Measured by Hospital Anxiety and Depression (HADS) Score (Baseline vs Week 12)
Description: To assess the change from baseline of CNS toxicity as measured by Hospital Anxiety and Depression (HADS) score (baseline vs week 12)
Time Frame: baseline to week 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 5 months
Description: From date of informed consent to date of follow up visit
Arm/Group | Single Arm
Serious Adverse Events (participants affected / at risk) | 4/40
Other Adverse Events (participants affected / at risk) | 8/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=40)
Thombosed haemorrhoids (Blood and lymphatic system disorders) | 1 (1)
Deliberate overdose (Psychiatric disorders) | 1 (1)
Peripheral neuropathy (Nervous system disorders) | 1 (1)
Groin pain (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=40)
Bilateral Arm Pain (Musculoskeletal and connective tissue disorders) | 1
Ichthyosis (Skin and subcutaneous tissue disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal Colic (Renal and urinary disorders) | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Night Sweats (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No